CLINICAL TRIAL: NCT01197430
Title: Vertical Stability Training Effects on the Eye-Hand Coordination of Female Volleyball Players
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Physical Education College (Other)
Responsible Party: Chang Gung Memory Hospital
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 980035
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: volleyball; neck vertical stability training; eye-hand coordination
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: exercise training

SUMMARY:
Purpose: Optimal eye-hand coordination is important for volleyball players. Neck disorder may affect neck function and subsequently eye-hand coordination. The purpose of this study is to explore the vertical stability training effects on coordination of the upper extremities of female volleyball players.

Methods: This study surveyed 25 players of a volleyball team, randomly assigned into the group A (training 1st) and group B (training 2nd). The group A includes 13 volleyball players and the group B includes 12. Eye-hand coordination was tested by a self-developed hand-stroking table device and stay time and motion time of upper extremities were determined. There are two testing modes, regular and random. Motion time for the electric probe moving between target sensor and stay time for the electric probe staying on a target sensors were collected for each mode, before each session of training and after the end of the 2nd session. In the 1st session of training, group A started vertical stability training and group B did control training for six weeks. In the 2nd session of training, the training programs were shifted between group A and B for another six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female Volleyball Players

Exclusion Criteria:

* can't party in training

Ages: 17 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)